CLINICAL TRIAL: NCT01657227
Title: Effectiveness and Cost-effectiveness of Two Multi-component Interventions to Improve the Health Outcomes in People With Type 2 Diabetes Mellitus
Brief Title: Tertiary Prevention in Type II Diabetes Mellitus in Canary Islands Study
Acronym: INDICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Servicio Canario de Salud (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Asociación para la Diabetes de Tenerife (Unknown); Asociación de Diabéticos de Gran Canaria (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ADE10 00032
Record Dates: First submitted 2012-07-31; First posted 2012-08-06 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; self-management; lifestyle; diet; physical exercise; computer-assisted decision support systems
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participating FCUs were not told about their intervention assignment (groups 1-4) until the last patient agreed to participate at every FCU. To warrant patient participation and cooperation, interventions could neither be blinded to patients nor to healthcare professionals. Data analysis is blinded to the intervention assignment.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention to Patients (Experimental): Only patients receive intervention
  Interventions: Behavioral: Intervention to patients; Other: Usual care
- Intervention to healthcare Professionals (Experimental): Primary care physicians and nurses practitioners receive the intervention. Their associated patients do not receive direct intervention although indirect intervention through professionals
  Interventions: Behavioral: Intervention to professionals; Other: Usual care
- Mixed Intervention (Experimental): Patients and healthcare professionals (primary care physicians and nurses practitioners) associated with these patients receive intervention
  Interventions: Behavioral: Intervention to patients; Behavioral: Intervention to professionals; Other: Usual care
- Control (Other): Patients receive usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Intervention to patients — Multifaceted intervention consisting of:
  * Program of education and behavior modification: group sessions conducted by health educators for the patient and a relative (who usually do the food shopping or prepare meals) every 3 months over 2 years (total:8 sessions). Main contents: diabetes, hygiene/nutrition and physical exercise.
  * Monitoring of patient conditions by Informational Communication Technologies (ICT): patient will complete at home a web-based short questionnaire once a week and an expanded version once a month.
  * Short text messaging to patient's mobile based on information obtained from self-reported questionnaires. 3 types of messages: 1) Reminders for completing web-based questionnaires, the attendance at group sessions and the follow-up appointments, 2) General advice on good habits, 3) Custom messages to reinforce behavior change.
  Arms: Intervention to Patients; Mixed Intervention
Behavioral: Intervention to professionals — Multifaceted intervention consisting of:
  * Educational intervention: Two theoretical and practical sessions to update knowledge on T2DM management and provide professionals with techniques to enhance the patient-centered clinical relationship model and the shared decision making model with the ultimate goal of improving patient adherence to treatment and self-care.
  * Computer-based clinical decision support system (CDSS): Implementation of an automated tool combining evidence-based knowledge with patient-specific information to assist clinicians in making clinical decisions in the management of T2DM patients.
  * Feedback: periodic mailing of personalized feedback reports with data on health results of all T2DM patients who are cared by the professional.
  Arms: Intervention to healthcare Professionals; Mixed Intervention
Other: Usual care — Usual care for T2DM received in primary health care

SUMMARY:
Objective:

* To improve health outcomes of patients with type 2 diabetes mellitus (T2DM) by influencing disease self-management through lifestyle modification and by helping primary care professionals to improve health care provided to patients.
* To assess the effectiveness and cost-effectiveness of two complex interventions (education and behavioural modification, independently and conjointly, for primary health care teams (PHCT) and patients and their relatives) to improve the health results in people with T2DM.

Methodology:

Design: Randomized clinical trial. Setting: Basic healthcare district in Canary Islands. Spain. Subjects: Patients with T2DM, 18-65 years old, without complications. Main measures: HbA1c, rate of patients with properly controlled T2DM. Sample: 2328 patients, 582 per arm. Intervention: G1: Interventions on the patients: Educational and habit modification group program. G2: Intervention on the PHCT: a) Educative intervention to improve the knowledge about the disease and their abilities; b) Computer-based clinical decision support system; c) Feedback of results. G3: Interventions on the patients and the PHCT. G4: Control group. Patients receive only the usual care.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* T2DM diagnosis
* aged between 18 and 65

Health professionals:

* primary health care teams (PHCT) comprising a primary care physician and a nurse practitioner associated to a patient will be selected
* must have a permanent position or a stable substitute position

Exclusion Criteria:

* peripheral vascular disease
* diabetic nephropathy and/or chronic kidney disease
* cognitive impairment, dementia
* major depression
* insufficient level of Spanish
* to be pregnant or planning to become pregnant in the next 6 months
* cancer last 5 years
* ischemic disease or heart failure
* proliferative diabetic retinopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2334 (Actual)
Dates: Start 2013-01; Primary Completion 2016-10-20 (Actual); Study Completion 2016-10-20 (Actual)

PRIMARY OUTCOMES:
Change in Glycosylated hemoglobin (HbA1c) | Baseline and 12 months
  Change in Glycosylated hemoglobin from baseline to 12 months

SECONDARY OUTCOMES:
Change in Glycosylated hemoglobin (HbA1c) | Baseline and 3, 6, 18 and 24 months
Change in Weight | Baseline and 3, 6, 12, 18 and 24 months
Change in Waist circumference | Baseline and 3, 6, 12, 18 and 24 months
Change in Body Mass Index (BMI) | Baseline and 3, 6,12, 18 and 24m
Change in Basal glucose | Baseline and 3, 6, 12, 18 and 24 months
Change in Total cholesterol level | Baseline and 6, 12 and 24 months
Change in HDL level | Baseline and 6, 12 and 24 months
Change in LDL level | Baseline and 6, 12 and 24 months
Change in Triglycerides | Baseline and 6, 12 and 24 months
Change in EQ-5D index | Baseline and 6, 12, 18 and 24 months
  EQ-5D is a generic questionnaire for health related quality of life (HRQL) assessment
Change in ADDQoL score | Baseline and 6, 12, 18 and 24 months
  ADDQoL is a specific questionnaire for health related quality of life (HRQL) assessment
Medication administration | Baseline and 6, 12, 18 and 24 months
  Initiation of new drugs or dosage adjustment: insulin, antidiabetics, hypolipidemics, antihypertensives, etc.
Change in tabacco consumption | Baseline and 3, 6, 12, 18 and 24 months
Acceptability of interventions and satisfaction (INDICA-SATP) | 24 months
Change in Diabetes Knowledge | Baseline, 12 and 24 months
Change in Mediterranean Diet Adherence Screener (MEDAS) score | Baseline and 6, 12, 18 and 24 months
Change in International Physical Activity Questionnarie (IPAQ) score | Baseline and 6, 12, 18 and 24 months
Change in Stait-Trait Anxiety Inventory (STAI) score | Baseline, 12 and 24 months
Change in Beck Depression Inventory - II (BDI-II) score | Baseline, 12 and 24 months
Change in Diabetes Distress Scale (DDS2) score | Baseline, 12 and 24 months
Change in Diabetes Empowerment Scale - Short Form (DES-SF) score | Baseline, 12 and 24 months
Change in Morisky Compliance Scale | Baseline and 6, 12, 18 and 24 months

OTHER OUTCOMES:
Incidence of micro- and macrovascular complications | Baseline, 12 and 24 months
  Coronary events, peripheral vascular complications, cerebral vascular complications, diabetic retinopathy, diabetic nephropathy
Quality measures of the T2DM care process | Baseline and 6, 12, 18 and 24 months
  Adherence to recommendations on physical exam, lab test and treatment
Resource utilization and costs | Baseline and 3, 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pedro G Serrano-Aguilar, MD, PhD, Principal Investigator — Servicio de Evaluación del Servicio Canario de la Salud; Pedro Serrano Aguilar, MD, PhD, Study Director — Servicio de Evaluación del Servicio Canario de la Salud; Pedro Serrano Aguilar, MD, PhD, Study Chair — Servicio de Evaluación del Servicio Canario de la Salud
Locations (1):
- Servicio de Evaluación del Servicio Canario de la Salud, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia-Perez L, Ramallo-Farina Y, Vallejo-Torres L, Rodriguez-Rodriguez L, Gonzalez-Pacheco H, Santos-Hernandez B, Garcia-Bello MA, Wagner AM, Carmona M, Serrano-Aguilar PG; INDICA team. Cost-effectiveness of multicomponent interventions in type 2 diabetes mellitus in a cluster randomised controlled trial: the INDICA study. BMJ Open. 2022 Apr 8;12(4):e058049. doi: 10.1136/bmjopen-2021-058049. PMID 35396305
- [Derived] Ramallo-Farina Y, Rivero-Santana A, Garcia-Perez L, Garcia-Bello MA, Wagner AM, Gonzalez-Pacheco H, Rodriguez-Rodriguez L, Kaiser-Girardot S, Monzon-Monzon G, Guerra-Marrero C, Daranas-Aguilar C, Roldan-Ruano M, Carmona M, Serrano-Aguilar PG; INDICA Team. Patient-reported outcome measures for knowledge transfer and behaviour modification interventions in type 2 diabetes-the INDICA study: a multiarm cluster randomised controlled trial. BMJ Open. 2021 Dec 15;11(12):e050804. doi: 10.1136/bmjopen-2021-050804. PMID 34911711
- [Derived] Ramallo-Farina Y, Garcia-Bello MA, Garcia-Perez L, Boronat M, Wagner AM, Rodriguez-Rodriguez L, de Pablos-Velasco P, Llorente Gomez de Segura I, Gonzalez-Pacheco H, Carmona Rodriguez M, Serrano-Aguilar P; INDICA Team. Effectiveness of Internet-Based Multicomponent Interventions for Patients and Health Care Professionals to Improve Clinical Outcomes in Type 2 Diabetes Evaluated Through the INDICA Study: Multiarm Cluster Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Nov 2;8(11):e18922. doi: 10.2196/18922. PMID 33136059
- [Derived] Ramallo-Farina Y, Garcia-Perez L, Castilla-Rodriguez I, Perestelo-Perez L, Wagner AM, de Pablos-Velasco P, Dominguez AC, Cortes MB, Vallejo-Torres L, Ramirez ME, Martin PP, Garcia-Puente I, Salinero-Fort MA, Serrano-Aguilar PG; INDICA team. Effectiveness and cost-effectiveness of knowledge transfer and behavior modification interventions in type 2 diabetes mellitus patients--the INDICA study: a cluster randomized controlled trial. Implement Sci. 2015 Apr 9;10:47. doi: 10.1186/s13012-015-0233-1. PMID 25880498